CLINICAL TRIAL: NCT01412541
Title: A Prospective, Multicenter, Single Blind, Randomized, Controlled Trial Comparing the Moxy Drug Coated Balloon vs. Standard Balloon Angioplasty for Treatment of Femoropopliteal Arteries
Brief Title: Moxy Drug Coated Balloon vs. Standard Balloon Angioplasty for the Treatment of Femoropopliteal Arteries
Acronym: LEVANT 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL0002-01
Record Dates: First submitted 2011-08-05; First posted 2011-08-09 (Estimated); Results first posted 2016-03-29 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Femoral Artery Stenosis; Popliteal Artery Stenosis; Femoral Artery Occlusion; Popliteal Artery Occlusion
Keywords: Arms; Experimental; Drug Coated Angioplasty Balloon; Active Comparator; Standard Angioplasty Balloon
MeSH Terms: conditions — Rhabdomyosarcoma, Alveolar

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All Duplex Ultrasound operators, core lab evaluators, and members of the Clinical Events Committee (CEC) will be blinded to the subject's treatment assignment. Both the subject as well as the Investigator conducting the follow-up visit will be blinded to treatment until the completion of the 12 month visit.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moxy Drug Coated Balloon (Experimental): Paclitaxel coated balloon catheter
  Interventions: Device: Moxy Drug Coated Balloon
- Standard Uncoated Angioplasty Balloon (Active Comparator): PTA Catheter
  Interventions: Procedure: Standard Uncoated Angioplasty Balloon

INTERVENTIONS:
Procedure: Standard Uncoated Angioplasty Balloon — Subjects will be randomized 2:1 to the Moxy Drug Coated Balloon or Standard Angioplasty Balloon
  Arms: Standard Uncoated Angioplasty Balloon
Device: Moxy Drug Coated Balloon — Subjects will be randomized 2:1 to the drug coated or standard angioplasty balloon
  Arms: Moxy Drug Coated Balloon

SUMMARY:
The purpose of the study is to demonstrate the superior efficacy and non-inferior safety of the Moxy Drug Coated Balloon by direct comparison to standard percutaneous transluminal angioplasty (PTA) catheter for treatment of stenosis of the femoropopliteal arteries.

DETAILED DESCRIPTION:
The Moxy Drug Coated Balloon is indicated for percutaneous transluminal angioplasty of obstructive de novo or non-stented restenotic lesions in native femoropopliteal arteries up to 15 cm in length and ≥4.0 to ≤6.0 mm in diameter. This study will randomize approximately 476 patients who will receive either the Moxy balloon or standard balloon angioplasty at 55 global investigational sites. Subjects will be blinded to treatment until 12 months and will participate in long term follow-up for 5 years.

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Male or non-pregnant female ≥18 years of age;
2. Rutherford Clinical Category 2-4;
3. Patient is willing to provide informed consent, is geographically stable and comply with the required follow up visits, testing schedule and medication regimen;

   Angiographic Lesion Inclusion Criteria:
4. Length ≤15 cm;
5. Up to two focal lesions or segments within the designated 15 cm length of vessel may be treated (e.g. two discrete segments, separated by several cm, but both falling within a composite length of ≤15 cm);
6. ≥70% stenosis by visual estimate;
7. Lesion location starts ≥1 cm below the common femoral bifurcation and terminates distally ≤2 cm below the tibial plateau AND ≥1 cm above the origin of the TP trunk;
8. de novo lesion(s) or non-stented restenotic lesion(s) >90 days from prior angioplasty procedure;
9. Lesion is located at least 3 cm from any stent, if target vessel was previously stented;
10. Target vessel diameter between ≥4 and ≤6 mm and able to be treated with available device size matrix;
11. Successful, uncomplicated (without use of a crossing device) antegrade wire crossing of lesion;
12. A patent inflow artery free from significant lesion (≥50% stenosis) as confirmed by angiography (treatment of target lesion acceptable after successful treatment of inflow artery lesions); NOTE: Successful inflow artery treatment is defined as attainment of residual diameter stenosis ≤30% without death or major vascular complication.
13. At least one patent native outflow artery to the ankle, free from significant (≥50%) stenosis as confirmed by angiography that has not previously been revascularized (treatment of outflow disease is NOT permitted during the index procedure);
14. Contralateral limb lesion(s) cannot be treated within 2 weeks before and/or planned 30 days after the protocol treatment in order to avoid confounding complications;
15. No other prior vascular interventions within 2 weeks before and/or planned 30 days after the protocol treatment.

Exclusion Criteria:

Patients will be excluded if ANY of the following conditions apply:

1. Pregnant or planning on becoming pregnant or men intending to father children;
2. Life expectancy of <5 years;
3. Patient is currently participating in an investigational drug or other device study or previously enrolled in this study; NOTE: Enrollment in another clinical trial during the follow up period is not allowed.
4. History of hemorrhagic stroke within 3 months;
5. Previous or planned surgical or interventional procedure within 2 weeks before or within 30 days after the index procedure;
6. History of myocardial infarction (MI), thrombolysis or angina within 2 weeks of enrollment;
7. Rutherford Class 0, 1, 5 or 6;
8. Renal failure or chronic kidney disease with modification in diet in renal disease glomerular filtration rate (MDRD GFR) ≤30 ml/min per 1.73 m2 (or serum creatinine ≥2.5 mg/L within 30 days of index procedure or treated with dialysis);
9. Prior vascular surgery of the index limb, with the exception of remote common femoral patch angioplasty separated by at least 2 cm from the target lesion;
10. Inability to take required study medications or allergy to contrast that cannot be adequately managed with pre- and post-procedure medication;
11. Anticipated use of IIb/IIIa inhibitor prior to randomization;
12. Ipsilateral retrograde access;
13. Composite lesion length is >15 cm or there is no normal proximal arterial segment in which duplex flow velocity can be measured;
14. Significant inflow disease. Successful treatment of inflow disease allowed prior to target lesion treatment;
15. Known inadequate distal outflow (>50 % stenosis of distal popliteal and/or all three tibial vessels), or planned future treatment of vascular disease distal to the target lesion;
16. Sudden symptom onset, acute vessel occlusion, or acute or sub-acute thrombus in target vessel;
17. Severe calcification that renders the lesion un-dilatable;
18. Use of adjunctive treatment modalities (i.e. laser, atherectomy, cryoplasty, scoring/cutting balloon, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Rosenfield, MD, Principal Investigator — Massachusetts General Hospital; Prof. Dierk Scheinert, Principal Investigator — University Leipzig
Locations (54):
- United States (42):
  - Good Samaritan Hospital, Los Angeles, California
  - North County Radiology Medial Group Inc., Oceanside, California
  - St. Joseph's Hospital, Orange, California
  - University of California Davis, Sacramento, California
  - Medical Center of the Rockies, Loveland, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Washington Cardiology Center, Washington D.C., District of Columbia
  - Heart and Vascular Institute, Clearwater, Florida
  - Interventional Cardiolgists of Gainesville, Gainesville, Florida
  - Munroe Regional Medical Center, Ocala, Florida
  - Cardiovascular Associates, Elk Grove Village, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Edward Heart, Oakbrook Terrace, Illinois
  - St. John's Hospital, Springfield, Illinois
  - Allen County Cardiology, Fort Wayne, Indiana
  - St. Vincent Heart Center of Indianapolis, Indianapolis, Indiana
  - Methodist Medical Center, Des Moines, Iowa
  - Promise Regional Medical Center, Hutchinson, Kansas
  - St. Francis Heart & Vascular Center, Topeka, Kansas
  - Massachusetts Genearl Hospital, Boston, Massachusetts
  - Detroit Medical Center, Detroit, Michigan
  - St. John's Hospital, Detroit, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Mercy Hosptial, Coon Rapids, Minnesota
  - Forrest General Hospital, Hattiesburg, Mississippi
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Our Lady of Lourdes Medical Center, Cherry Hill, New Jersey
  - New York University Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia Universtiy Medical Center, New York, New York
  - Wake Heart and Vascular, Raleigh, North Carolina
  - Christ Hospital / The Lindner Clinical Trial Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Mid Ohio Cardiology and Vascular Consultants, Columbus, Ohio
  - Jobst Vascular Institute, Toledo, Ohio
  - Univesrity of Toledo Medical Center, Toledo, Ohio
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Wellmont Cardiology Services, Kingsport, Tennessee
  - East Tennessee Heart Consultants, Knoxville, Tennessee
  - Baptist DeSoto in Southaven, Memphis, Tennessee
  - Austin Heart P.A., Austin, Texas
- Austria (2):
  - Medical University of Graz, Graz
  - Medical University of Vienna, Vienna
- Belgium (2):
  - Imelda Ziekenhuis, Bonheiden
  - Flanders Medical Research Program, Dendermonde
- Germany (8):
  - Herz-Zentrum, Bad Krozingen
  - Jewish Hospital, Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Diakonissenanstalt zu Flensburg, Flensburg
  - Hamburg University Cardiovascular Center, Hamburg
  - University Leipzig, Leipzig
  - University Magdeburg, Magdeburg
  - University of Tübingen, Tübingen

REFERENCES:
- [Derived] Ouriel K, Adelman MA, Rosenfield K, Scheinert D, Brodmann M, Pena C, Geraghty P, Lee A, White R, Clair DG. Safety of Paclitaxel-Coated Balloon Angioplasty for Femoropopliteal Peripheral Artery Disease. JACC Cardiovasc Interv. 2019 Dec 23;12(24):2515-2524. doi: 10.1016/j.jcin.2019.08.025. Epub 2019 Sep 28. PMID 31575518
- [Derived] Scheinert D, Schmidt A, Zeller T, Muller-Hulsbeck S, Sixt S, Schroder H, Weiss N, Ketelsen D, Ricke J, Steiner S, Rosenfield K. German Center Subanalysis of the LEVANT 2 Global Randomized Study of the Lutonix Drug-Coated Balloon in the Treatment of Femoropopliteal Occlusive Disease. J Endovasc Ther. 2016 Jun;23(3):409-16. doi: 10.1177/1526602816644592. Epub 2016 Apr 26. PMID 27117972
- [Derived] Rosenfield K, Jaff MR, White CJ, Rocha-Singh K, Mena-Hurtado C, Metzger DC, Brodmann M, Pilger E, Zeller T, Krishnan P, Gammon R, Muller-Hulsbeck S, Nehler MR, Benenati JF, Scheinert D; LEVANT 2 Investigators. Trial of a Paclitaxel-Coated Balloon for Femoropopliteal Artery Disease. N Engl J Med. 2015 Jul 9;373(2):145-53. doi: 10.1056/NEJMoa1406235. Epub 2015 Jun 24. PMID 26106946

RESULTS

PARTICIPANT FLOW:
Groups:
- Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB): Test group: Formerly called the Moxy Drug Coated Balloon, the Lutonix DCB is a paclitaxel coated balloon catheter
  Subjects were randomized 2:1 to the Lutonix DCB or standard angioplasty balloon.
- Standard Uncoated Angioplasty Balloon: Control group: standard uncoated PTA catheter
  Subjects were randomized 2:1 to the Lutonix DCB or standard angioplasty balloon.
Period: Overall Study
Arm/Group | Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) | Standard Uncoated Angioplasty Balloon
Started | 372 | 160
Completed | 246 | 117
Not Completed | 126 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) | Standard Uncoated Angioplasty Balloon | Total
Number analyzed (Participants) | 372 | 160 | 532
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (10.0) | 69.0 (9.0) | 68.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 53 | 198
  Male | 227 | 107 | 334

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Composite Freedom From All-Cause Peri-Operative (≤30 Day) Death and Freedom From Index Limb Amputation, Index Limb Re-Intervention, and Index-Limb-Related Death at 12 Months Post Index Procedure
Description: Composite of freedom from all-cause peri-operative (≤30 day) death and freedom at 1 year from the following: index limb amputation (above or below the ankle), index limb re-intervention, and index-limb-related death.
Time Frame: 12 months post index procedure
Population: The number of participants (n) varies from the total number of participants (N) in the study as n depends on the number of participants for which data was available at the given time-point analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 335 | 146
Percentage of participants | 85.4 [81.6 to 89.2] | 79.5 [72.9 to 86.0]
Statistical Analysis 1: Comparison: Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) vs Standard Uncoated Angioplasty Balloon; To assess if proportion of subjects with at least one safety event* in the Test group is inferior or not inferior to that of Control group through 12-months Post index procedure (PPI) H0: The proportion of subjects with safety events in the Test group through 12-months PPI is clinically inferior to that of the Control group. H1: The proportion of subjects with safety events in the Test group through 12-months PPI is clinically non-inferior to that of the Control group; Test type: Non-Inferiority or Equivalence — The evaluable sample size required for 90% power is 150 (50 Control plus 100 Test). This endpoint is not the sample-size driver of the study. Randomization of 476 subjects is expected to provide at least 405 evaluable subjects, after adjustment for up to 15% censoring) and approximately 99% power; p = 0.025, Farrington and Manning

2. Primary Outcome: Percentage of Participants With Primary Patency of the Target Lesion at 12 Months Post Index Procedure
Description: Primary Patency is defined as the absence of target lesion restenosis (defined by DUS peak systolic velocity ratio (PSVR) ≥2.5) and freedom from target lesion revascularization (TLR).
Time Frame: 12 months post index procedure
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 314 | 137
Percentage of participants | 66.6 [61.3 to 71.8] | 54.0 [45.7 to 62.4]
Statistical Analysis 1: Comparison: Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) vs Standard Uncoated Angioplasty Balloon; To assess whether the proportion of subjects with at least one efficacy event* in the Test group is equal or not to that of Control group through 12-months post-index procedure. H0: The proportion of subjects with efficacy events in the Control group through 12-months post-index procedure is equal to that of the Test group. H1: The proportion of subjects with efficacy events in the Control group through 12-months post-index procedure is not equal to that of the Test group; Test type: Equivalence — The statistical analysis is a likelihood ratio chi-square test for inequality of binomial proportions; the test is a two-sided test at α=0.05. The response variable in each subject will be the presence or absence of at least one efficacy event from the time following the index procedure through 12 months. The study evaluable sample size required for 90% power is approximately 405 subjects. After adjustment for 15% censoring through 12 months, the study size is 476; p = 0.05, Chi-squared; The statistical analysis is a likelihood ratio chi-square test for inequality of binomial proportions; the test is a two-sided test

3. Secondary Outcome: Number of Acute Device Success at Time of Index Procedure
Description: Device Success was defined as the achievement of successful delivery and deployment of the study device(s) as intended at the intended target lesion, without balloon rupture or inflation/deflation abnormalities and a successful withdrawal of the study system.
Time Frame: At time of Index Procedure
Population: as for outcome 1
Measure: Count of Units; unit: Devices
Units Other Than Participants: Devices
Arm/Group | Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 372 | 160
Number analyzed (Devices) | 432 | 180
Devices | 430 | 180

4. Secondary Outcome: Number of Participants With Technical and Procedural Success
Description: Technical Success is defined as successful access and deployment of the device and visual estimate of ≤30% diameter residual stenosis during the index procedure without deployment of a bailout stent.
  Procedural Success is defined as attainment of ≤30% residual stenosis in the treatment area by independent core lab analysis without serious adverse events during the index procedure.
Time Frame: At time of Index Procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 372 | 160
Participants
  Technical Success | 282 | 138
  Procedural Success | 281 | 138

5. Secondary Outcome: Number of Participants With Primary Patency at 6, 12, and 24 Months Post Index Procedure
Description: Primary Patency is defined as the absence of target lesion restenosis (defined by core lab adjudication or strict application of PSVR thresholds) and freedom from target lesion revascularization (TLR).
Time Frame: 6, 12, and 24 months post index procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 372 | 160
Participants
  6 months post index procedure: number analyzed (Participants) | 326 | 142
  6 months post index procedure | 263 | 92
  12 months post index procedure: number analyzed (Participants) | 314 | 137
  12 months post index procedure | 209 | 74
  24 months post index procedure: number analyzed (Participants) | 294 | 127
  24 months post index procedure | 160 | 60

6. Secondary Outcome: Number of Participants With Alternative Primary Patency at 6, 12, and 24 Months Post Index Procedure
Description: Percentage of subjects with Alternative Primary Patency based on alternative definitions of duplex ultrasound (DUS) peak systolic velocity ratio (PSVR) <2.0 and <3.0 at 6, 12, and 24 months post index procedure. DUS PSVR was calculated by dividing the maximum peak systolic velocity (PSV) from the stenosis by the PSV from the nearest segment of normal artery above the site of increase.
Time Frame: 6, 12, and 24 months post index procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 372 | 160
Participants
  DUS PSVR <2.0 : 6 months post index procedure: number analyzed (Participants) | 314 | 135
  DUS PSVR <2.0 : 6 months post index procedure | 220 | 74
  DUS PSVR <2.0 : 12 months post index procedure: number analyzed (Participants) | 296 | 133
  DUS PSVR <2.0 : 12 months post index procedure | 158 | 62
  DUS PSVR <2.0 : 24 months post index procdure: number analyzed (Participants) | 262 | 113
  DUS PSVR <2.0 : 24 months post index procdure | 106 | 38
  DUS PSVR <3.0 : 6 months post index procedure: number analyzed (Participants) | 313 | 136
  DUS PSVR <3.0 : 6 months post index procedure | 259 | 98
  DUS PSVR <3.0 : 12 months post index procedure: number analyzed (Participants) | 286 | 127
  DUS PSVR <3.0 : 12 months post index procedure | 197 | 73
  DUS PSVR <3.0 : 24 months post index procdure: number analyzed (Participants) | 244 | 105
  DUS PSVR <3.0 : 24 months post index procdure | 131 | 48

7. Secondary Outcome: Number of Participants With Duplex Ultrasound (DUS) Clinical Patency at 6, 12, and 24 Months Post Index Procedure
Description: DUS Clinical Patency defined as DUS PSVR <2.5 without prior clinically driven target lesion revascularization (TLR).
Time Frame: 6, 12, and 24 months post index porcedure
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 372 | 160
Participants
  6 months post index procedure: number analyzed (Participants) | 312 | 137
  6 months post index procedure | 252 | 90
  12 months post index procedure: number analyzed (Participants) | 288 | 130
  12 months post index procedure | 188 | 69
  24 months post index procedure: number analyzed (Participants) | 249 | 107
  24 months post index procedure | 123 | 42

8. Secondary Outcome: Number of Participants With Freedom From Target Lesion Revascularization (TLR) Clinically-driven at 6, 12, and 24 Months Post Index Procedure
Time Frame: 6, 12, and 24 months post index procedure
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 372 | 160
Participants
  6 months post index procedure: number analyzed (Participants) | 349 | 153
  6 months post index procedure | 329 | 144
  12 months post index procedure: number analyzed (Participants) | 334 | 146
  12 months post index procedure | 296 | 122
  24 months post index procedure: number analyzed (Participants) | 309 | 138
  24 months post index procedure | 250 | 104

9. Secondary Outcome: Improvement in Rutherford Classification Scores at 6, 12, and 24 Months Post Index Procedure Compared to Baseline
Description: The endpoint summarizes the change in index-limb Rutherford Classification of participants from baseline through 24 months. Data is presented as shift from baseline Rutherford Classification data using the following categories: 1) Improvement, 2) Same, and 3) Worsened.
Time Frame: 6, 12, and 24 months post index procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Moxy Drug Coated Balloon | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 372 | 160
Participants
  6 months from baseline: number analyzed (Participants) | 333 | 145
  6 months from baseline: Improved | 290 | 118
  6 months from baseline: Same | 30 | 22
  6 months from baseline: Worsened | 13 | 5
  12 months from baseline: number analyzed (Participants) | 309 | 131
  12 months from baseline: Improved | 273 | 108
  12 months from baseline: Same | 27 | 21
  12 months from baseline: Worsened | 9 | 2
  24 months from baseline: number analyzed (Participants) | 280 | 122
  24 months from baseline: Improved | 242 | 106
  24 months from baseline: Same | 31 | 15
  24 months from baseline: Worsened | 7 | 1

10. Secondary Outcome: Change in Resting Ankle Brachial Index (ABI) at 6, 12, and 24 Months Compared to Baseline
Description: Mean change from baseline values. The Ankle Brachial Index (ABI) is defined as a ratio of ankle to brachial (upper arm) artery systolic blood pressure and aims at determining how well the blood is flowing in the legs.
Time Frame: 6, 12, and 24 months from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 372 | 160
Index
  6 months post index procedure: number analyzed (Participants) | 320 | 135
  6 months post index procedure | 0.20 (0.24) | 0.16 (0.22)
  12 months post index procedure: number analyzed (Participants) | 300 | 126
  12 months post index procedure | 0.18 (0.24) | 0.18 (0.25)
  24 months post index procedure: number analyzed (Participants) | 269 | 112
  24 months post index procedure | 0.14 (0.27) | 0.17 (0.24)

11. Secondary Outcome: Change in Six Minute Walk Test Distance at 6, 12, and 24 Months Compared to Baseline
Description: The data bellow is presented as a Mean change in scores for the Six Minute Walk Test scores at 6, 12, and 24 months compared to baseline.
Time Frame: 6, 12, and 24 months from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 372 | 160
Meters
  6 months from baseline: number analyzed (Participants) | 265 | 131
  6 months from baseline | 42.5 (205.7) | 61.1 (213.4)
  12 months from baseline: number analyzed (Participants) | 244 | 120
  12 months from baseline | 45.0 (227.5) | 37.4 (120)
  24 months from baseline: number analyzed (Participants) | 217 | 104
  24 months from baseline | 48.6 (190.6) | 47.1 (209.2)

12. Secondary Outcome: Change in European Quality of Life 5 Dimensions (EuroQol -5D) Scores at 6, 12, and 24 Months Compared to Baseline.
Description: Mean change in EuroQol (EQ-5D) scores at 6, 12, and 24 months compared to baseline. The EurolQol-5D system rates quality of life using five dimensions including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels of ratings, that is, no problems, slight problems, moderate problems, severe problems and extreme problems that can be selected. A visual scale allows participants to report their own perception of their health status. The overall scores range from 0 (worst) to 100 (best). Please note that the data in the table below represent the mean changes in overall scores for each group compared to their baseline data.
Time Frame: 6, 12, and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 372 | 160
Score on a scale
  6 months from baseline: number analyzed (Participants) | 265 | 137
  6 months from baseline | 0.08 (0.21) | 0.10 (0.18)
  12 months from baseline: number analyzed (Participants) | 250 | 127
  12 months from baseline | 0.09 (0.20) | 0.08 (0.20)
  24 months from baseline: number analyzed (Participants) | 222 | 120
  24 months from baseline | 0.07 (0.23) | 0.09 (0.20)

13. Secondary Outcome: Change in Score on the Short Form Quality of Life Measure (Physical Component) at 6, 12, and 24 Months Compared to Baseline.
Description: Mean change from Baseline on the Short Form (SF-36 v2) Quality of Life Questionnaire at 6, 12, and 24 months. The SF-36 v2 United States (US) is a brief measure of general health status. The physical health measure of the test comprises four scales, that is, physical functioning (10 items), role-physical (4 items), bodily pain (2 items), and general health (5 items). The scores range between 0 and 100 (with higher scores indicating better health). In the results presented below, a positive Mean represents an increase in the average health score while a negative Mean represents a decrease in the same mean score compared to baseline measure.
Time Frame: 6, 12, and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 372 | 160
score on a scale
  6 months from baseline: number analyzed (Participants) | 286 | 142
  6 months from baseline | 6.6 (11.4) | 6.3 (10.0)
  12 months from baseline: number analyzed (Participants) | 263 | 133
  12 months from baseline | 6.0 (11.4) | 5.4 (10.2)
  24 months from baseline: number analyzed (Participants) | 240 | 122
  24 months from baseline | 4.5 (11.2) | 5.2 (9.9)

14. Secondary Outcome: Change in Quality of Life (Mental Component) on the Short-form 36 (SF-36 v2) at 6, 12, and 24 Months Compared to Baseline
Description: Mean change in quality of life (mental component) on Short-form 36 (SF-36 v2) from baseline at 6, 12, and 24 months. The SF-36 v2 United States (US) is a brief measure of general health status. The mental health measure comprises four scales, that is, vitality (4 items), social functioning (2 items), role-emotional (3 items), and mental health (5 items). The scores range from 0 to 100 (with higher scores indicating better health). In the results presented below, a positive Mean represents an increase in the average health score while a negative Mean represents a decrease in the same mean score compared to baseline measure.
Time Frame: 6, 12, and 24 months from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 372 | 160
score on a scale
  6 months from baseline: number analyzed (Participants) | 286 | 142
  6 months from baseline | -0.7 (12.0) | 1.6 (14.1)
  12 months from baseline: number analyzed (Participants) | 263 | 133
  12 months from baseline | 0.2 (12.4) | 0.4 (13.4)
  24 months from baseline: number analyzed (Participants) | 240 | 122
  24 months from baseline | -0.4 (13.0) | 1.8 (13.5)

15. Secondary Outcome: Number of Subjects With Freedom From Death, Index-Limb Amputation, and Target Vessel Revascularization (TVR) at 30 Days Post Index Porcedure
Description: Number of subjects with Freedom from all-cause death, index limb amputation above the ankle and Target Vessel Revascularization (TVR) (VIVA Safety Endpoint)
Time Frame: 30 days post index procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Lutonix 035 Drug Coated Balloon (Lutonix DCB): Test group: Formerly called the Moxy Drug Coated Balloon, the Lutonix DCB is a paclitaxel coated balloon catheter
  Subjects were randomized 2:1 to the Lutonix DCB or standard angioplasty balloon.
Arm/Group | Lutonix 035 Drug Coated Balloon (Lutonix DCB) | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 362 | 156
Participants | 361 | 155

16. Secondary Outcome: Number of Participants With Composite of Freedom From All-Cause Perioperative (<30 Day) Death and Freedom From the Following at 1,6, 24, 36, 48, and 60 Months: Index Limb Amputation, Index Limb Re-intervention, and Index Limb Related Death
Time Frame: 1, 6, 24, 36, 48, and 60 months post index procedure
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 372 | 160
Participants
  1 month post index procedure: number analyzed (Participants) | 362 | 156
  1 month post index procedure | 360 | 155
  6 months post index procedure: number analyzed (Participants) | 350 | 153
  6 months post index procedure | 324 | 140
  24 months post index procedure: number analyzed (Participants) | 310 | 140
  24 months post index procedure | 240 | 94
  36 months post index procedure: number analyzed (Participants) | 294 | 137
  36 months post index procedure | 212 | 87
  48 months post index procedure: number analyzed (Participants) | 281 | 133
  48 months post index procedure | 189 | 74
  60 months post index procedure: number analyzed (Participants) | 260 | 129
  60 months post index procedure | 160 | 69

17. Secondary Outcome: Number of Participants With All Cause Death, Amputation, Target Vessel Revascularization, Reintervention for Thrombosis, Major and Minor Vascular Complications, and Readmission for Cardiovascular Events at 1, 6, 12, 24, 36, 48, and 60 Months PPI.
Description: Amputation defined as above the ankle free survival (AFS). PPI = Post index procedure.
Time Frame: 1, 6, 12, 24, 36, 48, and 60 months post index procedure
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 372 | 160
participants
  Death : 1 month PPI: number analyzed (Participants) | 362 | 156
  Death : 1 month PPI | 0 | 0
  Death : 6 months PPI: number analyzed (Participants) | 354 | 154
  Death : 6 months PPI | 4 | 2
  Death : 12 months PPI: number analyzed (Participants) | 341 | 148
  Death : 12 months PPI | 10 | 4
  Death : 24 months PPI: number analyzed (Participants) | 326 | 141
  Death : 24 months PPI | 25 | 8
  Death : 36 months PPI: number analyzed (Participants) | 320 | 139
  Death : 36 months PPI | 37 | 10
  Death : 48 months PPI: number analyzed (Participants) | 316 | 137
  Death : 48 months PPI | 54 | 14
  Death : 60 months PPI: number analyzed (Participants) | 306 | 133
  Death : 60 months PPI | 64 | 17
  Major Amputation : 1 month PPI: number analyzed (Participants) | 362 | 156
  Major Amputation : 1 month PPI | 0 | 0
  Major Amputation : 6 months PPI: number analyzed (Participants) | 350 | 153
  Major Amputation : 6 months PPI | 1 | 0
  Major Amputation : 12 months PPI: number analyzed (Participants) | 335 | 144
  Major Amputation : 12 months PPI | 1 | 0
  Major Amputation : 24 months PPI: number analyzed (Participants) | 305 | 134
  Major Amputation : 24 months PPI | 1 | 0
  Major Amputation : 36 months PPI: number analyzed (Participants) | 286 | 131
  Major Amputation : 36 months PPI | 1 | 0
  Major Amputation : 48 months PPI: number analyzed (Participants) | 267 | 124
  Major Amputation : 48 months PPI | 2 | 1
  Major Amputation : 60 months PPI: number analyzed (Participants) | 245 | 116
  Major Amputation : 60 months PPI | 2 | 1
  Minor Amputation : 1 month PPI: number analyzed (Participants) | 362 | 156
  Minor Amputation : 1 month PPI | 0 | 0
  Minor Amputation : 6 months PPI: number analyzed (Participants) | 349 | 153
  Minor Amputation : 6 months PPI | 0 | 0
  Minor Amputation : 12 months PPI: number analyzed (Participants) | 334 | 144
  Minor Amputation : 12 months PPI | 0 | 0
  Minor Amputation : 24 months PPI: number analyzed (Participants) | 304 | 134
  Minor Amputation : 24 months PPI | 1 | 0
  Minor Amputation : 36 months PPI: number analyzed (Participants) | 285 | 131
  Minor Amputation : 36 months PPI | 2 | 0
  Minor Amputation : 48 months PPI: number analyzed (Participants) | 267 | 124
  Minor Amputation : 48 months PPI | 3 | 0
  Minor Amputation : 60 months PPI: number analyzed (Participants) | 244 | 116
  Minor Amputation : 60 months PPI | 3 | 0
  Amputation Free Survival : 1 month PPI: number analyzed (Participants) | 362 | 156
  Amputation Free Survival : 1 month PPI | 362 | 156
  Amputation Free Survival : 6 months PPI: number analyzed (Participants) | 353 | 154
  Amputation Free Survival : 6 months PPI | 349 | 152
  Amputation Free Survival : 12 months PPI: number analyzed (Participants) | 341 | 148
  Amputation Free Survival : 12 months PPI | 331 | 144
  Amputation Free Survival : 24 months PPI: number analyzed (Participants) | 326 | 141
  Amputation Free Survival : 24 months PPI | 301 | 133
  Amputation Free Survival : 36 months PPI: number analyzed (Participants) | 320 | 139
  Amputation Free Survival : 36 months PPI | 283 | 129
  Amputation Free Survival : 48 months PPI: number analyzed (Participants) | 316 | 137
  Amputation Free Survival : 48 months PPI | 261 | 122
  Amputation Free Survival : 60 months PPI: number analyzed (Participants) | 306 | 133
  Amputation Free Survival : 60 months PPI | 242 | 115
  Total TLR : 1 month PPI: number analyzed (Participants) | 362 | 156
  Total TLR : 1 month PPI | 1 | 0
  Total TLR : 6 months PPI: number analyzed (Participants) | 349 | 153
  Total TLR : 6 months PPI | 20 | 9
  Total TLR : 12 months PPI: number analyzed (Participants) | 334 | 146
  Total TLR : 12 months PPI | 38 | 24
  Total TLR : 24 months PPI: number analyzed (Participants) | 309 | 138
  Total TLR : 24 months PPI | 59 | 34
  Total TLR : 36 months PPI: number analyzed (Participants) | 292 | 135
  Total TLR : 36 months PPI | 69 | 38
  Total TLR : 48 months PPI: number analyzed (Participants) | 278 | 130
  Total TLR : 48 months PPI | 78 | 45
  Total TLR : 60 months PPI: number analyzed (Participants) | 256 | 126
  Total TLR : 60 months PPI | 85 | 46
  Total TVR : 1 month PPI: number analyzed (Participants) | 362 | 156
  Total TVR : 1 month PPI | 1 | 1
  Total TVR : 6 months PPI: number analyzed (Participants) | 349 | 153
  Total TVR : 6 months PPI | 22 | 12
  Total TVR : 12 months PPI: number analyzed (Participants) | 334 | 146
  Total TVR : 12 months PPI | 42 | 26
  Total TVR : 24 months PPI: number analyzed (Participants) | 309 | 138
  Total TVR : 24 months PPI | 63 | 39
  Total TVR : 36 months PPI: number analyzed (Participants) | 292 | 135
  Total TVR : 36 months PPI | 73 | 43
  Total TVR : 48 months PPI: number analyzed (Participants) | 278 | 130
  Total TVR : 48 months PPI | 83 | 53
  Total TVR : 60 months PPI: number analyzed (Participants) | 256 | 126
  Total TVR : 60 months PPI | 90 | 54
  Reintervention for Thrombosis : 1 month PPI: number analyzed (Participants) | 362 | 156
  Reintervention for Thrombosis : 1 month PPI | 1 | 1
  Reintervention for Thrombosis : 6 months PPI: number analyzed (Participants) | 349 | 153
  Reintervention for Thrombosis : 6 months PPI | 1 | 1
  Reintervention for Thrombosis : 12 months PPI: number analyzed (Participants) | 334 | 144
  Reintervention for Thrombosis : 12 months PPI | 1 | 1
  Reintervention for Thrombosis : 24 months PPI: number analyzed (Participants) | 304 | 134
  Reintervention for Thrombosis : 24 months PPI | 1 | 1
  Reintervention for Thrombosis : 36 months PPI: number analyzed (Participants) | 285 | 131
  Reintervention for Thrombosis : 36 months PPI | 2 | 1
  Reintervention for Thrombosis : 48 months PPI: number analyzed (Participants) | 266 | 124
  Reintervention for Thrombosis : 48 months PPI | 2 | 1
  Reintervention for Thrombosis : 60 months PPI: number analyzed (Participants) | 243 | 116
  Reintervention for Thrombosis : 60 months PPI | 2 | 1
  Cardiovascular Hospitalization : 1 month PPI: number analyzed (Participants) | 362 | 156
  Cardiovascular Hospitalization : 1 month PPI | 1 | 0
  Cardiovascular Hospitalization : 6 months PPI: number analyzed (Participants) | 349 | 153
  Cardiovascular Hospitalization : 6 months PPI | 20 | 3
  Cardiovascular Hospitalization : 12 months PPI: number analyzed (Participants) | 334 | 144
  Cardiovascular Hospitalization : 12 months PPI | 31 | 10
  Cardiovascular Hospitalization : 24 months PPI: number analyzed (Participants) | 308 | 135
  Cardiovascular Hospitalization : 24 months PPI | 52 | 21
  Cardiovascular Hospitalization : 36 months PPI: number analyzed (Participants) | 293 | 132
  Cardiovascular Hospitalization : 36 months PPI | 55 | 23
  Cardiovascular Hospitalization : 48 months PPI: number analyzed (Participants) | 279 | 126
  Cardiovascular Hospitalization : 48 months PPI | 55 | 23
  Cardiovascular Hospitalization : 60 months PPI: number analyzed (Participants) | 262 | 119
  Cardiovascular Hospitalization : 60 months PPI | 55 | 23
  Major Vascular Complication : 1 month PPI: number analyzed (Participants) | 362 | 156
  Major Vascular Complication : 1 month PPI | 15 | 2
  Major Vascular Complication : 6 months PPI: number analyzed (Participants) | 350 | 153
  Major Vascular Complication : 6 months PPI | 19 | 4
  Major Vascular Complication : 12 months PPI: number analyzed (Participants) | 335 | 145
  Major Vascular Complication : 12 months PPI | 22 | 7
  Major Vascular Complication : 24 months PPI: number analyzed (Participants) | 310 | 135
  Major Vascular Complication : 24 months PPI | 32 | 10
  Major Vascular Complication : 36 months PPI: number analyzed (Participants) | 294 | 132
  Major Vascular Complication : 36 months PPI | 36 | 13
  Major Vascular Complication : 48 months PPI: number analyzed (Participants) | 282 | 126
  Major Vascular Complication : 48 months PPI | 39 | 13
  Major Vascular Complication : 60 months PPI: number analyzed (Participants) | 263 | 119
  Major Vascular Complication : 60 months PPI | 39 | 13

18. Secondary Outcome: Change in Walking Impairment Questionnaire (WIQ) Scores at 6, 12, and 24 Months Post Index Procedure Compared to Baseline.
Description: The WIQ assesses 3 categories of activities that include 1) walking distance, 2) stair-climbing, and 3) walking speed. Each question requires participants to rate their degree of difficulty with the activity on a scale of 0 (unable) to 4 (no problem). Final scores range from 0% to 100%, with lower percentages indicating higher levels of difficulties with activities.The results below represent the mean differences in total Walking Impairment Questionnaire (WIQ) scores at 6, 12, and 24 months, compared to baseline assessment scores.
Time Frame: 6, 12, and 24 months post index procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lutonix 035 Drug Coated Balloon PTA Catheter (Lutonix DCB) | Standard Uncoated Angioplasty Balloon
Number analyzed (Participants) | 372 | 160
score on a scale
  6 months from baseline: number analyzed (Participants) | 280 | 134
  6 months from baseline | 26.6 (28.8) | 20.5 (28.7)
  12 months from baseline: number analyzed (Participants) | 261 | 130
  12 months from baseline | 23.9 (27.6) | 19.2 (26.5)
  24 months from baseline: number analyzed (Participants) | 236 | 122
  24 months from baseline | 22.4 (28.8) | 16.9 (26.7)

ADVERSE EVENTS:
Time Frame: 60 months
Description: All adverse events occurring in this study will be classified in accordance with the adverse event signs or symptoms.
  Both Non-Serious Adverse Events (AE) and Serious Adverse Events (SAE) are reported with a threshold of 3%.
Arm/Group | Lutonix 035 Drug Coated Balloon (Lutonix DCB) | Standard Uncoated Angioplasty Balloon
All-Cause Mortality (participants affected / at risk) | 64/372 | 17/160
Serious Adverse Events (participants affected / at risk) | 289/372 | 125/160
Other Adverse Events (participants affected / at risk) | 316/372 | 126/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lutonix 035 Drug Coated Balloon (Lutonix DCB) (N=372) | Standard Uncoated Angioplasty Balloon (N=160)
Angina, stable (Cardiac disorders) | 28 | 8
Angina, Unstable (Cardiac disorders) | 10 | 5
Arrhytmia, Other (Cardiac disorders) | 14 | 10
Chronic heart failure (Cardiac disorders) | 18 | 8
Hypertension (Cardiac disorders) | 10 | 10
Myocardial infarction (Cardiac disorders) | 24 | 17
Cardiovascular, Other (Cardiac disorders) | 59 | 20
Diarrhea (Gastrointestinal disorders) | 2 | 6
Gastrointestinal bleeding (Gastrointestinal disorders) | 20 | 8
Gastrointestinal, Others (Gastrointestinal disorders) | 22 | 11
Local infection (Infections and infestations) | 8 | 8
Stroke -ischemic (Nervous system disorders) | 15 | 3
Other neurological - nervous system (Nervous system disorders) | 15 | 7
Carcinoma (Respiratory, thoracic and mediastinal disorders) | 12 | 3
Other respiratory (Respiratory, thoracic and mediastinal disorders) | 21 | 6
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 32 | 7
Fracture (bone) (Musculoskeletal and connective tissue disorders) | 13 | 10
Claudication (Musculoskeletal and connective tissue disorders) | 3 | 6
Other skeletal, spine and muscular system (Musculoskeletal and connective tissue disorders) | 32 | 12
Restenosis (Vascular disorders) | 65 | 33
Occlusion/closure (Vascular disorders) | 6 | 5
Restenosis (Vascular disorders) | 19 | 18
Renal failure/ insufficiency (Renal and urinary disorders) | 20 | 9
Urinary infection (Renal and urinary disorders) | 8 | 5
Other genito-urinary system (Renal and urinary disorders) | 10 | 5
Carcinoma (General disorders) | 26 | 5
Other (General disorders) | 65 | 21
Arterial occlusion (Vascular disorders) | 12 | 9
Atherosclerosis (Vascular disorders) | 15 | 11
Restenosis (Vascular disorders) | 32 | 22
Stenosis (Vascular disorders) | 42 | 23
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lutonix 035 Drug Coated Balloon (Lutonix DCB) (N=372) | Standard Uncoated Angioplasty Balloon (N=160)
Hematoma bleeding puncture site minor (General disorders) | 23 | 4
Angina, Stable (Vascular disorders) | 23 | 11
Angina, Unstable (Vascular disorders) | 12 | 2
Arrythmia - other (Cardiac disorders) | 13 | 10
Hypertension (Vascular disorders) | 21 | 9
Hypotension (Vascular disorders) | 13 | 3
Other - Cardiovascular (Vascular disorders) | 43 | 23
Diabetes Melitus Type II (Endocrine disorders) | 12 | 7
Nausea (Gastrointestinal disorders) | 13 | 2
Other- gastrointestinal (Gastrointestinal disorders) | 39 | 11
Infection, local (Infections and infestations) | 20 | 12
Other infectious (Infections and infestations) | 12 | 4
Dizziness/ vertigo (Nervous system disorders) | 19 | 9
Other neurological/ nervous system (Nervous system disorders) | 38 | 13
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 22 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 24 | 7
Other respiratory (Respiratory, thoracic and mediastinal disorders) | 36 | 18
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 16 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 14 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 45 | 8
Fracture (bone) (Musculoskeletal and connective tissue disorders) | 17 | 7
Claudication (Musculoskeletal and connective tissue disorders) | 24 | 17
Other skeletal, spine and muscular system (Musculoskeletal and connective tissue disorders) | 117 | 35
Dissection (General disorders) | 11 | 6
Restenosis (Vascular disorders) | 18 | 11
Restenosis in target vessel (Vascular disorders) | 14 | 3
Renal failure/ insufficiency (Renal and urinary disorders) | 22 | 5
Urinary infection (Renal and urinary disorders) | 26 | 9
Other, genito-urinary system (Renal and urinary disorders) | 24 | 13
Rash (Skin and subcutaneous tissue disorders) | 12 | 5
Other (General disorders) | 157 | 67
Restenosis (Vascular disorders) | 13 | 3
Stenosis (Vascular disorders) | 15 | 5
Other vessel specific (Vascular disorders) | 14 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-03-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT01412541/Prot_SAP_000.pdf